CLINICAL TRIAL: NCT00136110
Title: A Randomized, Double-Blind, Placebo-Controlled Sequential Clinical Trial of Sodium Valproate in ALS
Brief Title: Trial of Sodium Valproate in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/182-0
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2007-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Sodium Valproate; randomised trial; Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Valproic Acid

INTERVENTIONS:
Drug: Sodium Valproate

SUMMARY:
The purpose of this study is to determine whether the use of sodium valproate is effective in slowing the disease progression in Amyotrophic Lateral Sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a devastating disease characterized by progressive degeneration of motor neurons leading to muscle weakness.

The pathogenesis of ALS is unknown, but there is convincing evidence that several molecular mechanisms play a role. Previous studies investigated the role of the Survival Motor Neuron (SMN) gene in ALS. Recent data suggest that SMN genotypes producing less SMN protein increase susceptibility and severity of ALS. This leads to the hypothesis that the clinical expression of ALS is influenced by the total SMN protein level in affected patients. In a population of ALS patients in the Netherlands we found that SMN genotypes producing less SMN protein appear to increase susceptibility and severity of ALS. It was shown that the HDAC inhibitor sodium valproate (SVP) increases levels of SMN protein in vitro. From these results and from data suggesting neuroprotective properties of SVP, it is hypothesised that SVP could extend survival of patients with ALS. In addition, sodium valproate significantly prolonged the disease duration in the animal model for ALS, the SOD1 transgenic mouse. Given that SVP is a FDA-approved compound with well-known pharmacokinetic and toxicity profiles, it is an attractive candidate for a clinical trial in ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Definite, probable, or probable-laboratory supported ALS according to the revised El Escorial World Federation of Neurology criteria.
* Intake of riluzole 50 mg twice a day (bid)
* A disease duration at inclusion of more than 6 months and less than 36 months [inclusive] (disease onset is defined as the date of first symptoms excluding muscle cramps and fasciculations)
* Vital capacity (VC%) ≥ 70% of normal value (slow expiration, best of a minimum of three and a maximum of five measurements, with a respiratory function validly assessable and a spontaneous, non-assisted ventilation)
* Ages 18 - 85 years (inclusive)
* Capable of thoroughly understanding the trial information given; has signed the informed consent.

Exclusion Criteria:

* Tracheostomy, tracheostomal ventilation of any type, non-invasive ventilation more than 16 hours/ day, or supplemental oxygen during the last three months prior to inclusion.
* Any medical condition or intoxication known to have an association with motor neuron dysfunction, which might confound or obscure the diagnosis of ALS.
* Presence of any concomitant life-threatening disease or any disease or impairment likely to interfere with functional assessment.
* Confirmed hepatic insufficiency or abnormal liver function (ASAT, ALAT greater than twice the upper limit of normal range).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-04; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
The rate of decline of daily functioning

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Van den Berg, MD, PhD, Study Chair — UMC Utrecht; Sanne Piepers, MD, Principal Investigator — UMC Utrecht; Sonja W De Jong, MD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Piepers S, Veldink JH, de Jong SW, van der Tweel I, van der Pol WL, Uijtendaal EV, Schelhaas HJ, Scheffer H, de Visser M, de Jong JM, Wokke JH, Groeneveld GJ, van den Berg LH. Randomized sequential trial of valproic acid in amyotrophic lateral sclerosis. Ann Neurol. 2009 Aug;66(2):227-34. doi: 10.1002/ana.21620. PMID 19743466